CLINICAL TRIAL: NCT04033666
Title: Comparative Analysis of Non-invasive Ventilatory Support Modes: High Flow Nasal Cannula and Non-invasive Ventilation in Acute Asthmatic Children
Brief Title: Analysis of Non-invasive Ventilatory Support Modes: High Flow Nasal Cannula and Non-invasive Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Evelim Leal de Freitas Dantas Gomes, PT, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: High Flow Nasal Cannula
Record Dates: First submitted 2019-07-12; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Asthma Acute
Keywords: asthma; High flow nasal cannula; Non invasive ventilation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial comparing high-flow nasal cannula intervention with non-invasive ventilation with two levels of pressure in children hospitalized for acute asthma
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome accessor and the investigator when evaluating the child and the spreadsheet data will not know which therapy the patient was submitted to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow nasal cannula (Active Comparator): It will be administered as part of the high-flow nasal cannula treatment to reduce the symptoms of acute asthma
  Interventions: Other: High Flow Nasal cannula
- NIV noninvasive ventilation (Active Comparator): It will be administered as part of the Noninvasive ventilation treatment to reduce the symptoms of acute asthma
  Interventions: Other: NIV Noninvasive Ventilation

INTERVENTIONS:
Other: High Flow Nasal cannula — The HFNC will be instituted therapy with high-flow nasal cannula with dosage and cannula calculated according to the child's weight, ranging from 2 l / min to 30 l / min. The therapy will begin with diaphragmatic exercises 3x10 breaths and after high-flow therapy with nasal cannula for 45 minutes, after which will be performed the vital signs evaluations and Peak Flow, HRV, FEV1.
  Other Names: HFNC
  Arms: High Flow nasal cannula
Other: NIV Noninvasive Ventilation — The Therapy consisted of 3x10 diaphragmatic re-education exercises after a Bipap device was coupled in bipedal mode with parameters Ipap 12 cm H2O and Epap 8 cm H2O, for 45 minutes, according to the patient's tolerance, with Full face facial mask. After therapy evaluated vital signs and measures of Peak Flow, HRV, FEV1.
  Other Names: NIV
  Arms: NIV noninvasive ventilation

SUMMARY:
This study compares two types of noninvasive treatments for asthma attacks with the objective of analyzing the efficacy of each therapy during the period of exacerbations in infants and asthmatics hospitalized.

DETAILED DESCRIPTION:
A randomized clinical trial, where it will be established, treatment in hospitalized asthma patients in the infirmary and Emergency Room of the Hospital Infantil Cândido Fontoura.

The children eligible for the Protocol, after signing the terms of consent and assent, will be randomized for treatment in 2 groups (GI - bilevel and GII - High Flow Nasal Cannula). After the evaluations are started: Feb1, Volume expired in the first second; Peak Flow, vital signs and calculated Pulmonary Asthma Score, Pulmonary Asthma Severity Score, Pulmonary Index Score, and therapy application. The N to be considered for the study of 20 individuals per group. Group therapy I will be applied in diaphragmatic re-education exercises 3 x 10 breaths, after non-invasive ventilation, with parameters 12 cm H2O Ipap and Epap 8 cm H2O, for 45 minutes, according to patient tolerance, interface, with full face mask After treatment, reassessment of vital signs and measurements of Peak Flow, Fev1 and Severity Scores.

The GII will be established therapy with high-flow nasal cannula with dosage and cannula calculated according to the child's weight and respiratory rate at the time of evaluation, ranging from 2 l / min to 30 l / min. flow. The therapy will begin with diaphragmatic exercises 3 x 10 breaths, after 45 minutes of the installation of the therapy that is continuous, will be performed a reassessment of vital signs and Peak Flow, Feb, Severity Scores.

During the hospitalization time of the child will be carried out the daily treatment, therapy chosen for each patient for 45 minutes in the case of GI and the GII group daily follow-up and adjustment of flow dosage, also evaluated the vital signs, vital signs and Peak Flow, Feb, Gravity Scores.

At the time of hospital discharge, the evaluations will be performed and data such as inhaled corticosteroid use, oxygen use in days and inspired fraction, hospitalization days, hospital costs, as well as vital signs, vital signs and Peak Flow, Fev, Scores of Gravity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 16 years;
* both genders;
* Be in the presence of the bronchospasm crisis;
* Be admitted to HICF Hospital;
* Have signed the search terms

Exclusion Criteria:

* Having associated heart disease;
* neurological/cognitive impairment;
* Have severe respiratory insufficiency detected by severity scores;
* Intolerance to any type of treatment

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
PAS Pediatric Asthma Score | Change from baseline PAS at first 45 minutes and 5th day in hospital
  PAS Pediatric Asthma Score- This score assesses respiratory distress and wheezing. Higher score the more severe the asthma attack. The score ranges from 3 to 15 and clinical improvement is expected when there is a reduction of 3 points or more.
Suplemental Oxigen day use | Change from baseline Oxygen dose at first 45 minutes and 5th day in hospital.
  Oxigen dose number of days used

SECONDARY OUTCOMES:
Forced Expiratory volume in first second | Change from baseline FEV1 at first 45 minutes and 5th day in hospital.
  FEV1 liters and percentage
Bronchodilator doses ( Salbutamol) | Change from baseline Salbutamol dose (First day and 5th day in hospital)
  Amount of puffs administered per day

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Costa, Principal Investigator — University of Nove de Julho
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] David MMC, Gomes ELFD, Cavassini CLF, Luiz JG, Costa D. Comparison of the effects of high-flow nasal cannula and bilevel positive airway pressure treatments as respiratory physiotherapy interventions for children with asthma exacerbation: a randomized clinical trial. Einstein (Sao Paulo). 2024 Aug 26;22:eAO0588. doi: 10.31744/einstein_journal/2024AO0588. eCollection 2024. PMID 39194097